CLINICAL TRIAL: NCT00214422
Title: A Pilot Study of Image Guided Prostate and Pelvic Nodal Irradiation With Intensity Modulated Radiation Therapy (IMRT) in Prostate Cancer
Brief Title: Intensity Modulated Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050241; 05-C-0241; NCT00278356 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2005-09-21 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; Radiation; Cancer; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1- 5040cGy to the lymph nodes (Experimental): 5040Gray (cGy) to the lymph nodes
  Interventions: Radiation: Radiation
- Arm 2 - 5400cGy to the lymph nodes (Experimental): 5400Gray (cGy) to the lymph nodes
  Interventions: Radiation: Radiation
- Arm 3 - 5900cGy to the lymph nodes (Experimental): 5900Gray (cGy) to the lymph nodes
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.

SUMMARY:
BACKGROUND:

-This study represents a progression from findings in four previous National Cancer Institute (NCI) Radiation Oncology Branch (ROB) protocols (02-C-0167A, 02-C-0207E, 03-C-0190B, 04-C-0171). In these previous works we have begun to develop techniques to obtain Magnetic Resonance (MR) biological images and co-register tissue in prostate cancer patients.

OBJECTIVES:

-The primary objective of the first portion of this study is to assess the feasibility of using Intensity-modulated radiation therapy (IMRT) to treat the at-risk lymph nodes in prostate cancer. Also, if feasible, we hope optimize this technique with experience.

ELIGIBILITY:

-This is a study of image guided, targeted radiation therapy in patients with high risk of nodal metastases from prostate cancer. Patients with prostate cancer who have more than 15% risk of lymph node (as defined by the Partin tables) metastasis will be eligible for this study.

DESIGN:

* On the first 10 patients, we will perform approximately 5 computed tomography (CT) simulations throughout the course of their therapy. On each simulation, the initial treatment plan will be re-run. The dose-volume data from target and normal tissues will then be re-analyzed. From this analysis we will be better able to determine the size of margins needed to account for organ motion and changes such as varying amounts of gas in the bowel and fluid in the bladder. To the best of our knowledge, no such analyses have been published.
* If the initial part of this trial is feasible, we will proceed to a phase I dose escalation trial of radiation to the at-risk lymph nodes. The primary statistical objective of the phase I portion of this study is to estimate the Maximum Tolerated Dose (MTD) of external beam radiation based on evaluating acute toxicity. The study will be conducted with a dose-escalation design with 3 patients in each dose cohort. If fewer than 2 of 3 patients experience an acute dose limiting toxicity (DLT) than patients will be accrued to the next dose cohort. If 2 or more of 3 patients experience a DLT then the MTD will be exceeded and the prior, lower dose cohort will be considered the MTD. Secondary objectives of this study are to relate patterns in gene and protein expression to response and toxicity and to evaluate the frequency of late term toxicity.
* Specific procedures and risks will be described in a separate consent to be obtained at the time of biopsy. Tissue samples will be processed for complementary deoxyribonucleic acid (cDNA) microarray testing and stored for future analysis in the Radiation Oncology Branch, NCI.
* Anatomic Magnetic Resonance Imaging (MRI) and magnetic resonance (MR) biological images of the prostate and pelvis will be obtained and tissue will be acquired with biopsy locations precisely translated (co-registered) to an MR image of reference. A fiducial marker (gold seed) will be left at the biopsy site as a fiducial marker to direct future radiation therapy to the prostate. If necessary, additional fiducial markers will be placed for prostate localization during treatment.

DETAILED DESCRIPTION:
BACKGROUND:

-This study represents a progression from findings in four previous National Cancer Institute (NCI) Radiation Oncology Branch (ROB) protocols (02-C-0167A, 02-C-0207E, 03-C-0190B, 04-C-0171). In these previous works we have begun to develop techniques to obtain Magnetic Resonance (MR) biological images and co-register tissue in prostate cancer patients.

OBJECTIVES:

-The primary objective of the first portion of this study is to assess the feasibility of using Intensity-modulated radiation therapy (IMRT) to treat the at-risk lymph nodes in prostate cancer. Also, if feasible, we hope optimize this technique with experience.

ELIGIBILITY:

* This is a study of image guided, targeted radiation therapy in patients with high risk of nodal metastases from prostate cancer.
* Patients with prostate cancer who have more than 15% risk of lymph node (as defined by the Partin tables) metastasis will be eligible for this study.

DESIGN:

* On the first 10 patients, we will perform approximately 5 computed tomography (CT) simulations throughout the course of their therapy. On each simulation, the initial treatment plan will be re-run. The dose-volume data from target and normal tissues will then be re-analyzed. From this analysis we will be better able to determine the size of margins needed to account for organ motion and changes such as varying amounts of gas in the bowel and fluid in the bladder. To the best of our knowledge, no such analyses have been published.
* If the initial part of this trial is feasible, we will proceed to a phase I dose escalation trial of radiation to the at-risk lymph nodes. The primary statistical objective of the phase I portion of this study is to estimate the Maximum Tolerated Dose (MTD) of external beam radiation based on evaluating acute toxicity. The study will be conducted with a dose-escalation design with 3 patients in each dose cohort. If fewer than 2 of 3 patients experience an acute dose limiting toxicity (DLT) than patients will be accrued to the next dose cohort. If 2 or more of 3 patients experience a DLT then the MTD will be exceeded and the prior, lower dose cohort will be considered the MTD. Secondary objectives of this study are to relate patterns in gene and protein expression to response and toxicity and to evaluate the frequency of late term toxicity.
* Specific procedures and risks will be described in a separate consent to be obtained at the time of biopsy. Tissue samples will be processed for complementary deoxyribonucleic acid (cDNA) microarray testing and stored for future analysis in the Radiation Oncology Branch, NCI.
* Anatomic Magnetic Resonance Imaging (MRI) and magnetic resonance (MR) biological images of the prostate and pelvis will be obtained and tissue will be acquired with biopsy locations precisely translated (co-registered) to an MR image of reference. A fiducial marker (gold seed) will be left at the biopsy site as a fiducial marker to direct future radiation therapy to the prostate. If necessary, additional fiducial markers will be placed for prostate localization during treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Pathology report confirming adenocarcinoma of the prostate

Risk of lymph node metastasis greater than or equal to15% as defined by the Partin tables or biopsy proven positive lymph nodes

Tumor visible on magnetic resonance imaging (MRI)

No prior surgery, radiation, or chemotherapy for prostate cancer, with the exception of hormone therapy which may be given neoadjuvantly for up to four (4) months.

Age greater than 18 years old and less than 90 years old.

EXCLUSION CRITERIA:

Cognitively impaired patients who cannot give informed consent.

Patients with metastatic disease beyond the pelvis

Contraindication to biopsy

* Bleeding disorder
* Prothrombin time (PT)/partial thromboplastin time (PTT) greater than or equal to 1.5 times the upper limit of normal
* Platelets less than or equal to 50K
* Artificial heart valve

Contraindication to MRI

* Patients weighing greater than136 kgs (weight limit for the scanner tables)
* Allergy to magnetic resonance (MR) contrast agent
* Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices.

Pre-existing and active prostatitis or proctitis

Other medical conditions deemed by the principal investigator (PI) or associates to make the patient ineligible for protocol investigations, procedures, and high-dose external beam radiotherapy.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-09-19 (Actual); Primary Completion 2014-05-27 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Roach M 3rd, DeSilvio M, Lawton C, Uhl V, Machtay M, Seider MJ, Rotman M, Jones C, Asbell SO, Valicenti RK, Han S, Thomas CR Jr, Shipley WS; Radiation Therapy Oncology Group 9413. Phase III trial comparing whole-pelvic versus prostate-only radiotherapy and neoadjuvant versus adjuvant combined androgen suppression: Radiation Therapy Oncology Group 9413. J Clin Oncol. 2003 May 15;21(10):1904-11. doi: 10.1200/JCO.2003.05.004. PMID 12743142

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants in Arm 1 participated in a feasibility phase prior to the dose escalation phase of the study.
Groups:
- Arm 1- 5040cGy to the Lymph Nodes: 5040 Gray (cGy) to the lymph nodes
  Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.
- Arm 2 - 5400cGy to the Lymph Nodes: 5400cGy to the lymph nodes
  Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.
- Arm 3 - 5900cGy to the Lymph Nodes: 5900cGy to the lymph nodes
  Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.
Period: Overall Study
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGy to the Lymph Nodes
Started | 12 | 3 | 4
Completed | 7 | 2 | 3
Not Completed | 5 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Developed esophageal ca | 1 | 0 | 0
Not completed — Pt taken off study | 1 | 1 | 0
Not completed — Disease progression on study | 1 | 0 | 0
Not completed — Unable to make a radiation treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGy to the Lymph Nodes | Total
Number analyzed (Participants) | 12 | 3 | 4 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 0 | 9
  >=65 years | 5 | 1 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.14 (7.41) | 59.37 (20.36) | 67.68 (2.78) | 64.13 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 12 | 3 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 3 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 9 | 1 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 3 | 4 | 19
Median Prostatic Specific Antigen (PSA) at Diagnosis [Median (Full Range); unit: ng/ml] — Normal PSA is less than 2.5 ng/ml.
  ng/ml | 16.65 [5.5 to 103] | 33.4 [5.7 to 42.9] | 8.95 [4.75 to 27.3] | 19.67 [4.75 to 103]
Median Gleason Score at Diagnosis [Median (Full Range); unit: scores on a scale] — Gleason grading scale helps to evaluate the severity of prostate cancer. A score >8 is a low-grade cancer (less aggressive). A score <8 is a high grade cancer (more aggressive, poor prognosis).
  scores on a scale | 8 [7 to 9] | 7 [6 to 9] | 8 [7 to 8] | 7.6 [6 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Grade 2 Toxicity Using Intensity Modulated Radiation Therapy (IMRT) to Treat the At-risk Lymph Nodes in Prostate Cancer ( up to First 10 Patients)
Description: Radiation side effects were assessed by the Radiation Oncology Group (RTOG) Acute/Late Toxicity Grading Gastrointestinal and Genitourinary criteria. Acute Grade 0 - no symptoms, Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life threatening, and Grade 5 is death directly related to radiation side effects. Late toxicity is defined as occurring after 90 days.
Time Frame: At one week, one month, 2 months, 3 months, 6 months, 9 months, 1 year, 18 months, 2 years, 30 months, and 3 years after radiation therapy
Population: 6 participants in Arm 1 participated in a feasibility phase prior to the dose escalation phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes
Number analyzed (Participants) | 6
Participants
  Week 1 | 5
  1 month | 3
  2 months | 4
  3 months | 2
  6 months | 3
  9 months | 4
  1 year | 2
  18 months | 0
  2 years | 3
  30 months | 1
  3 years | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of External Beam Radiation to Pelvic Lymph Nodes of Interest in Patients Receiving Radiation Therapy for Prostate Cancer (After the First 10 Patients) In Arm 1, Arm 2, and Arm 3
Description: Maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 or more in a cohort of either 3 or 6 patients experiences a dose limiting toxicity (DLT) attributed to radiation therapy. An acute DLT will be defined as Radiation Therapy Oncology Group (RTOG) grade 3 or greater, acute gastrointestinal or genitourinary toxicity within 3 months after the completion of radiation.
Time Frame: Completion of Treatment, an average of 8.5 weeks
Population: The MTD of this study was not reached. The original principal investigator left the National Institutes of Health and we are unable to determine why the outcome was not met.
Groups:
- Arm 2 - 5400cGy to the Lymph Nodes; Arm 3 - 5900cGY to the Lymph Nodes: Radiation will be given in dose escalations from 5040 Gray (cGY) to a maximum of 5900 cGy to lymph nodes.
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGY to the Lymph Nodes
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Grade 2 Late Gastrointestinal or Genitourinary Toxicity Assessed by the Radiation Oncology Group (RTOG) Criteria
Description: Long-term effects and toxicity following intensity modulated radiation therapy (IMRT) dose escalation to the pelvic nodes were measured by the Radiation Oncology Group (RTOG) Criteria. Lower GI/Pelvis grade 2 toxicity Diarrhea requiring parasympatholytic drugs (e.g. Lomotil)/mucous discharge not necessitating sanitary pads/rectal or abdominal pain requiring analgesics and Genitourinary grade 2 defined as Frequency of urination or nocturia that is less frequent than every hour. Dysuria, urgency, bladder spasm requiring local anesthetic (e.g. Pyridium).
Time Frame: At median follow-up, approximately 28 months following radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGy to the Lymph Nodes
Number analyzed (Participants) | 12 | 3 | 4
Participants
  Gastrointestinal | 1 | 0 | 0
  Genitourinary | 3 | 0 | 0

4. Secondary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: An acute Dose Limiting Toxicity (DLT) will be defined as Radiation Therapy Oncology Group (RTOG) grade 3 or greater, acute gastrointestinal or genitourinary toxicity within 3 months after the completion of radiation.
Time Frame: Within 3 months after completion of radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGy to the Lymph Nodes
Number analyzed (Participants) | 12 | 3 | 4
Participants
  Gastrointestinal | 1 | 1 | 0
  Genitourinary | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 8 years and 3.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGy to the Lymph Nodes
Number analyzed (Participants) | 12 | 3 | 4
Participants | 12 | 3 | 4

6. Secondary Outcome: Number of Participants With Grade 3 or 4 Acute and/or Late Gastrointestinal or Genitourinary Toxicity Assessed by the Radiation Oncology Group (RTOG) Criteria
Description: Long-term effects and toxicity following intensity modulated radiation therapy (IMRT) dose escalation to the pelvic nodes were measured by the Radiation Oncology Group (RTOG) Criteria. Grade 3 toxicity Lower GI/Pelvis is Diarrhea requiring parenteral support/severe mucous or blood discharge necessitating sanitary pads/abdominal distention (flat plate radiograph demonstrates distended bowel loops), Grade 3 toxicity Genitourinary Frequency with urgency and nocturia hourly or more frequently/dysuria, pelvis pain or bladder spasm requiring regular, frequent narcotic/gross hematuria with/without clot passage.
Time Frame: At median follow-up, approximately 28 months following radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGY to the Lymph Nodes
Number analyzed (Participants) | 12 | 3 | 4
Participants
  Gastrointestinal | 1 | 1 | 0
  Genitourinary | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 8 years and 3.5 months.
Groups:
- Arm 1- 5040cGy to the Lymph Nodes: 5040 Gray (cGy) to the lymph nodes
  External Beam Radiation: Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.
- Arm 2 - 5400cGy to the Lymph Nodes: 5400cGy to the lymph nodes
  External Beam Radiation: Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.
- Arm 3 - 5900cGy to the Lymph Nodes: 5900cGy to the lymph nodes
  External Beam Radiation: Radiation will be given in dose escalations from 5040 Gray (cGy) to a maximum of 5900 cGy to lymph nodes.
Arm/Group | Arm 1- 5040cGy to the Lymph Nodes | Arm 2 - 5400cGy to the Lymph Nodes | Arm 3 - 5900cGy to the Lymph Nodes
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- 5040cGy to the Lymph Nodes (N=12) | Arm 2 - 5400cGy to the Lymph Nodes (N=3) | Arm 3 - 5900cGy to the Lymph Nodes (N=4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Liver (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- 5040cGy to the Lymph Nodes (N=12) | Arm 2 - 5400cGy to the Lymph Nodes (N=3) | Arm 3 - 5900cGy to the Lymph Nodes (N=4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Penis mass) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 8 (8) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 10 (16) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2)
Gastrointestinal - Other (Anal lesion - HPV virus (Bx on 1/28/18)) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (Diarrhea) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (Diarrhea, mucous discharge, abdo pain) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (Esophageal cancer) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (Urgency, abdominal pain) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (dysuria) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (frequency) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal - Other (increased bowel frequency) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (loose stools; frequency) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (mild BRBPR (hemorrhoids stable)) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (moderate diarrhea) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (moderate diarrhea, frequency, mucous) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (moderate frequency, urgency) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (rectal bleeding; urgency, frequent watery stools) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 0 (0)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (2)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 9 (20) | 3 (4) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Incontinence, anal (Gastrointestinal disorders) | 6 (9) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 4 (4) | 0 (0) | 1 (2)
Insomnia (General disorders) | 1 (2) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3)
Libido (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (3) | 4 (12)
Mood alteration::Depression (Nervous system disorders) | 3 (7) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Orgasmic dysfunction (Reproductive system and breast disorders) | 6 (6) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other (L shoulder) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other (R hip) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other (Thoracic back pain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 4 (6) | 1 (1) | 3 (4)
Pain::Breast (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pain::Pelvis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Dribbling) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Dysuria) (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (5)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 8 (10) | 2 (4) | 0 (0)
Weight gain (General disorders) | 10 (17) | 2 (3) | 0 (0)
Weight loss (General disorders) | 6 (8) | 1 (1) | 1 (1)
Cardiac General - Other (heart murmur) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Endocrine - Other (breast tenderness) (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal - Other (Incontinence) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other (blood streaked stool) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other (loose stool, urgency) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal - Other (loose stools) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal - Other (small amount blood in stools) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other (urgency) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint-function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Dysuria, Hematuria) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (nocturia) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Edema: limb (General disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine - Other (® thyroid size increased) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal - Other (frequency, soft BM's; mild abdo cramping) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 1 (2)
Hemorrhage, GU::Urethra (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Renal/Genitourinary - Other (Weak stream) (Renal and urinary disorders) | 6 (10) | 3 (4) | 1 (1)
Renal/Genitourinary - Other (dysuria, nocturia) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2011-07-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT00214422/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT00214422/Prot_SAP_001.pdf